CLINICAL TRIAL: NCT05324553
Title: Patient Derived Preclinical Models
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 21-008831
Record Dates: First submitted 2022-03-23; First posted 2022-04-12 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Cancer
Keywords: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Tissue Banks; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The collected tissue specimens will be used to develop preclinical models; i.e., cell lines, patient derived micro-cancer models as well as patient-derived xenograft models. In this study we may profile tumors using genomic and/or proteomic approaches to identify targetable alterations in tumor tissue from patients. To assure that the derived cell lines and micro-cancer models have not been cross contaminated during development with other models in development, DNA sequencing may be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Tissue Collection: Research tissue specimen will be obtained during the patient's clinical biopsy or clinical tumor resection, if feasible.
  Interventions: Procedure: Tissue Collection
- Blood Collection: Up to 50 mL of research blood will be drawn around the time of the procedure. Additional blood may be collected in selected cases, as warranted, to monitor disease recurrence/remission or perform additional testing
  Interventions: Diagnostic Test: Blood Collection
- Buccal Swab: Buccal swab may be requested, if necessary, to generate germline data.
  Interventions: Diagnostic Test: Buccal Swab

INTERVENTIONS:
Procedure: Tissue Collection — Research tissue specimen will be obtained during the patient's clinical biopsy or clinical tumor resection, if feasible.
  Groups: Tissue Collection
Diagnostic Test: Blood Collection — Up to 50 mL of research blood will be drawn around the time of the procedure. Additional blood may be collected in selected cases, as warranted, to monitor disease recurrence/remission or perform additional
  Groups: Blood Collection
Diagnostic Test: Buccal Swab — Buccal swab may be requested, if necessary, to generate germline data.
  Groups: Buccal Swab

SUMMARY:
Study goal is to collect tumor specimens that may inform cancer biology to eventually improve outcomes for patients with cancer. This proposal represents a highly collaborative effort to support cancer research with the goal of developing novel therapeutic strategies using patient derived preclinical models.

This study is being done to collect samples of tumor tissues, matched normal tissue when possible, and approximately 50 mL of blood.

DETAILED DESCRIPTION:
The objective of this study is to collect tumor specimens (tumor tissues, matched normal tissue when possible, and 50 mL of blood) that may inform cancer biology to eventually improve outcomes for patients with cancer. Additionally, relevant specimens that were previously collected under an IRB approved protocol (13-000942), will be used with approval of the PI of that protocol and patient consent for participation in this protocol.

The collected tissue specimens will be used to develop preclinical models; i.e., cell lines, patient derived micro-cancer models as well as patient-derived xenograft models. In this study we may profile tumors using genomic and/or proteomic approaches to identify targetable alterations in tumor tissue from patients. To assure that the derived cell lines and micro-cancer models have not been cross contaminated during development with other models in development, DNA sequencing may be used. Using these preclinical models, we will test new therapies in vitro, or in vivo in mice in order to identify novel therapeutics as well as interrogate genes for their role in tumor biology. Guidance for molecular targeted therapy will involve gene analysis of oncogenes and tumor suppressor genes. Results from these studies may provide the rationale for the design of future novel clinical trials. The evaluation of these preclinical models may lead to predictive value related to patient response to therapy as well as clinical trials. With consent, these models may be shared with other investigators internal or external to Mayo Clinic.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Patient is a good medical candidate for a standard of care or research biopsy or surgical procedure to obtain tissue

Exclusion Criteria:

* Uncontrolled concurrent illness including psychiatric illness, or situations that would limit compliance with the study requirements or the ability to willingly give written informed consent
* Institutionalized or incarcerated patients
* Inaccessible tumor for biopsy or patient does not have tumor tissue available for research use
* Biopsy must not be considered more than minimal risk to the patient.
* Have a contraindication to percutaneous biopsy including:

  1. Significant coagulopathy that cannot be adequately corrected.
  2. Severely compromised cardiopulmonary function or hemodynamic instability.
  3. Lack of a safe pathway to the lesion per the interventional radiologist.
  4. Inability of the patient to cooperate with, or to be positioned for, the procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient population includes anyone 18 years of age and older with cancer who are good medical candidates for standard of care or research biopsy or surgical procedure to obtain tissue.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-04-06 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants accrued with genomic, microbiome, and drug sensitivity components of aggressive cancer. | Up to 6 years post tissue and blood collection
  Sequencing data from DNA and RNA will be integrated into a visualization platform to allow individualized study of patient tumor mutations, rearrangements, and RNA expression. Genomically informed analysis will be employed to select potential targets for drug screening in the patient-derived 3D models and determine how many specimens are able to grow as 3D models. In some cases, immunostain results may be analyzed for correlation to RNA expression levels.

SECONDARY OUTCOMES:
Determine number of participants with genomic, microbiome and drug sensitivity assays (profile or functional) that suggest changes to treatment plan. | Up to 6 years post tissue and blood collection
  Sequencing data from DNA and RNA will be integrated into a visualization platform to allow individualized study of patient tumor mutations, rearrangements, and RNA expression. Genomically informed analysis will be employed to select potential targets for drug screening in the patient-derived 3D models. In some cases, immunostain results may be analyzed for correlation to RNA expression levels.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron S. Mansfield, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials